CLINICAL TRIAL: NCT06407830
Title: Effects of Motor Relearning Program With and Without Electrical Muscle Stimulation on Gait, Functional Independence and Quality of Life in Hemiplegic Stroke Patients
Brief Title: Effect of MRP With and Without EMS on Gait, Functional Independence and QOL in Stroke Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/23/0278
Record Dates: First submitted 2024-05-06; First posted 2024-05-09 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Stroke
Keywords: Gait; Functional independence; Quality of life
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention physical therapy (Active Comparator): Motor Relearning programme training
  Interventions: Other: motor relearning programme
- Electrical Muscle Stimulation (Experimental): Electrical Muscle Stimulation with Motor Relearning programme
  Interventions: Other: motor relearning programme; Other: electrical muscle stimulations with motor relearning programme

INTERVENTIONS:
Other: motor relearning programme — Treatment protocol includes Brief period of warm up and cool down (5 minutes). Individuals of this group will be provided 3 sessions per week; 1 hour per session; 24 sessions of task specific training based on the motor relearning programme. Each task specific training consists of 10 minutes.
Other: electrical muscle stimulations with motor relearning programme — Treatment protocol includes Brief period of warm up and cool down (5 minutes). Individuals of this group will be provided 3 sessions per week; 1 hour per session; 24 sessions of task specific training based on the motor relearning programme. Each task specific training consists of 10 minutes.
  Individuals of this group will be provided 3 sessions per week; 1 hour per session; 24 sessions for 8 weeks task specific training based on the motor relearning programme and 10 minutes of the EMS of each muscle during the session.
  Arms: Electrical Muscle Stimulation

SUMMARY:
To determine the effects of motor relearning programme with and without electrical muscle stimulation on gait, functional independence and quality of life in hemiplegic stroke patients.

DETAILED DESCRIPTION:
A study was performed a motor relearning program in stroke survivors. A clinically significant improvement was found in the motor relearning groups, and only in one study is this improvement significant compared to another intervention.

Neuromuscular Electrical Stimulation Improves Activities of Daily Living Post-Stroke. While the potential for enhancing functional motor ability seems less clear, the current systematic review and meta analysis's results point to a significant positive impact of NMES on ADL function during the post stroke rehabilitation process.

People with hemiparesis who received both conventional treatment and interventions based on motor relearning showed a significant improvement in their level of disability. There were no appreciable gains in the HRQoL perception.

Many research investigations have been carried out to assess the effects of motor relearning programs with regard to specific functional aspects and physical deficiencies. Up to the researcher's knowledge, there is no data to assess the effects of electrical muscle stimulation along with motor relearning programs in stroke patients. Therefore, the purpose of this study is to compare how a motor relearning program with and without electrical muscle stimulation affects hemiplegic stroke patients' gait, level of functional independence, and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed as hemiplegic stroke

  * Age between 45-65 years
  * Both males and females
  * Mini-Mental State Examination score ≥24
  * Able to stand independently for at least 1 min and (5) can ambulate 25 feet/10 m (with or without the assistive device)

Exclusion Criteria:

* Experiencing balance problems as a result of neurological conditions other than stroke (for instance cerebellar impairment, inner ear dysfunction, or Parkinson's disease)

  * Fixed ankle or foot contracture.
  * A serious cardiac disease (aorta stenosis, angina, hypertrophic cardiomyopathy, arrhythmia and pacemakers).
  * congenital limb deformities

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Functional Independence Measurement (FIM). | baseline week 1 and post interventional week 8
  The Functional Independence Measure (FIM) instrument was applied to assess the changes in functional ability. Out of the eighteen items in the FIM, thirteen evaluate physical domains and five evaluate cognitive functions. Each item is scored from 1 to 7 ("1" total dependence; "7" complete independence). The final score ranges from 18 to 126.

SECONDARY OUTCOMES:
Dynamic Gait Index | baseline week 1 and post interventional week 8
  The DGI has 8 items: walking, walking while changing speed, walking while turning the head horizontally and vertically, walking with pivot turn, walking over and around obstacles, and stair climbing. The scoring of the DGI is based on a 4-point scale ranging from 0 to 3, with 0 indicating severe impairment and 3 indicating normal ability. The best performance total score is 24. A low composite DGI score thus indicates greater impairment in functional mobility.
Stroke specific quality of life | baseline week 1 and post interventional week 8
  The SSQOL is a valid, reliable measurement that assesses health-related quality of life in stroke subjects and consists of a 49-item scale (each scored 1-5) representing 12 domains, for a maximum score of 245. All subjects were assessed while not wearing the treatment device.

CONTACTS AND LOCATIONS:
Overall Officials: Aruba Saeed, PhD, Principal Investigator — Riphah International University (Lahore)
Locations (1):
- Rehabilitation Center, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ghrouz A, Marco E, Munoz-Redondo E, Boza R, Ramirez-Fuentes C, Duarte E. The effect of motor relearning on balance, mobility and performance of activities of daily living among post-stroke patients: Study protocol for a randomised controlled trial. Eur Stroke J. 2022 Mar;7(1):76-84. doi: 10.1177/23969873211061027. Epub 2022 Feb 11. PMID 35300258
- [Background] Paolucci T, Agostini F, Mussomeli E, Cazzolla S, Conti M, Sarno F, Bernetti A, Paoloni M, Mangone M. A rehabilitative approach beyond the acute stroke event: a scoping review about functional recovery perspectives in the chronic hemiplegic patient. Front Neurol. 2023 Sep 15;14:1234205. doi: 10.3389/fneur.2023.1234205. eCollection 2023. PMID 37789885
- [Background] Mesci N, Ozdemir F, Kabayel DD, Tokuc B. The effects of neuromuscular electrical stimulation on clinical improvement in hemiplegic lower extremity rehabilitation in chronic stroke: a single-blind, randomised, controlled trial. Disabil Rehabil. 2009;31(24):2047-54. doi: 10.3109/09638280902893626. PMID 19874084